CLINICAL TRIAL: NCT05927844
Title: An Open, Single-arm, Multicenter Phase Ib Clinical Study of XH-30002 Capsule Combined With Afatinib Tablets for the Treatment of Locally Advanced or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: XH-30002 Capsule Combined With Afatinib Tablets for the Treatment of Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOG007
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Intervention Model Description: open, single-arm
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment ARM1 (Experimental): Drugs1：XH30002 Capsual 300mg，Qd，28d; Drug2：Afatiinb tablets 30mg，Qd，28d
  Interventions: Drug: XH-30002 capsule; Drug: Afatiinb tablet
- Treatment ARM2 (Experimental): Drugs1：XH30002 Capsual 400mg，Qd，28d; Drug2：Afatiinb tablets 30mg，Qd，28d
  Interventions: Drug: XH-30002 capsule; Drug: Afatiinb tablet

INTERVENTIONS:
Drug: XH-30002 capsule — receive the study drug until the investigator assessed no longer benefit, toxic intolerance, withdrawal of consent, loss of follow-up, or death, whichever occurred first
Drug: Afatiinb tablet — receive the study drug until the investigator assessed no longer benefit, toxic intolerance, withdrawal of consent, loss of follow-up, or death, whichever occurred first

SUMMARY:
This study is an exploratory clinical trial and does not involve statistical assumptions or sample size estimation. the mainly purpose for the study is to evaluate the safety of XH-30002 capsule combined with afatinib tablets in the treatment of locally advanced or metastatic esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This is an open, single-arm, multicenter, investigator-initiated Phase Ib clinical study to evaluate the efficacy and safety of XH-30002 capsule in combination with afatinib maleate tablets in patients with locally advanced or metastatic esophageal squamous cell carcinoma. The primary endpoint of the study was the safety of XH-30002 capsule combined with afatinib maleate tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study, agree to complete the corresponding visit and inspection according to the research plan, and sign the informed consent form (ICF);
2. Age ≥18 years old (as of the date of signing the ICF);
3. Esophageal squamous cell carcinoma confirmed by histology or cytology;
4. Patients with disease progression or intolerance after receiving at least first-line systemic treatment or refusing to accept standard treatment for various reasons;
5. The physical status score of the Eastern United States Oncology Consortium (ECOG) was 0-2;
6. Presence of at least one evaluable lesion according to RECIST 1.1 evaluation criteria;
7. Within 7 days before the first dose, the function of major organs and bone marrow meets the following criteria (in cases where blood transfusion or hematopoietic stimulation is not corrected within 14 days before the test) :

   1. Neutrophil count ≥1.5×109/L;
   2. Platelet count ≥100×109/L;
   3. Hemoglobin ≥90g/L;
   4. Liver function: For subjects with total bilirubin (TBIL) ≤1.5× upper reference value (ULN) or TBIL>1.5×ULN, direct bilirubin ≤1.0×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (liver metastasis subjects ≤5×ULN); Albumin ≥3.0g/dL;
   5. Renal function: serum creatinine ≤1.5×ULN or creatinine clearance ≥50mL/min (calculated by Cockcroft-Gault formula);
   6. Coagulation function: International standardized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5×ULN;
8. Expected survival time ≥3 months;
9. Women of reproductive age must undergo a negative blood pregnancy test within 7 days prior to enrollment and agree to use a reliable and effective method of contraception during the study treatment period and for 6 months after the last study treatment; For male subjects whose partner is a woman of reproductive age, consent must be given to use a reliable and effective method of contraception during the study treatment period and for 6 months after the last study treatment (whichever is the longest).

Exclusion Criteria:

1. Past or current use of afatinib maleate tablets or anti-tumor drugs targeting CDK4/6;
2. the presence of other active malignancies within 3 years prior to the first dose, except for locally curable tumors that have already received radical treatment (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, breast carcinoma in situ, early thyroid cancer, etc.);
3. Within 7 days before the first dose, there is uncontrollable serosal effusion requiring frequent drainage or medical intervention (such as pleural effusion, abdominal effusion, pericardial effusion, etc.);
4. Patients with central nervous system metastases (except asymptomatic brain metastases);
5. The toxicity level of previous anti-tumor therapy has not been restored to the General Adverse Event Term Standard 5.0 (CTCAE5.0) ≤ grade 1 (alopecia, peripheral neurotoxicity, simple laboratory tests and other toxicity that researchers judge no safety risk need to be mitigated to ≤ grade 2);
6. Those who have used potent inhibitors or inducers of CYP3A4 or CYP2C8 within 14 days before the first dose;
7. A history of hypersensitivity to any investigational drug ingredient or any known excipient
8. Patients with uncontrolled or significant cardiovascular and cerebrovascular diseases, including but not limited to:

   1. New York Heart Association (NYHA) Class II or higher congestive heart failure, unstable angina pectoris, myocardial infarction, or arrhythmia causing hemodynamic instability in the six months prior to screening;
   2. primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restricted cardiomyopathy, undefined cardiomyopathy);
   3. a history of clinically significant QT interval prolongation, or a screening period QTcF (calculated using Fridericia's formula) > 450 ms; Left ventricular ejection fraction (LVEF) ≤50%;
   4. Occurrence of arterial/venous thrombosis events, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc. within 6 months before screening;
9. Uncontrolled hypertension after optimal treatment (systolic blood pressure > 160mmHg or diastolic blood pressure > 100mmHg);
10. Esophagotracheal fistula, esophagomediastinal fistula, or tumor invasion risk of surrounding large blood vessels were diagnosed by imaging examination;
11. Gastrointestinal obstruction and active inflammatory bowel disease within 28 days prior to initial administration; The presence of chronic gastrointestinal dysfunction with diarrhea as the main symptom or other gastrointestinal disorders determined by investigators to be clinically significant, such as Crohn's disease, ulcerative colitis, malabsorption, or grade 1 diarrhea;
12. Patients with active hepatitis B [hepatitis B surface antigen (HBsAg) or HBcAb test positive and HBV-DNA≥ upper limit of normal] or hepatitis C [hepatitis C antibody (Anti-HCV) test positive and HCV-RNA≥ upper limit of normal] during the screening period;
13. Known history of human immunodeficiency virus (HIV) infection;
14. Serious chronic or active infected persons (including tuberculous infections) who require systemic antibacterial, antifungal, or antiviral treatment within 14 days prior to initial administration;
15. Received traditional Chinese medicine or radiation therapy with anti-tumor indications within 14 days before the first dose; Those who have received anti-tumor therapy such as targeted therapy, immunotherapy or other investigational drugs within 28 days or 5 half-lives prior to the first dose, whichever is shorter;
16. Those who had undergone major organ surgery within 28 days prior to initial dosing or planned to undergo elective surgery during the trial period (excluding needle biopsy);
17. Those who were vaccinated 28 days before the first dose or planned to be vaccinated during the trial;
18. Pregnant or lactating women;
19. Participating in other interventional clinical studies during the screening period (except non-interventional clinical studies or follow-up period of interventional studies);
20. Known history of mental or neurological disorders that may affect compliance with the test; People with drug or alcohol dependence; There are other investigators evaluating subjects who are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events and SAE | through study completion, an average of 6 months
  The Treatment-Related Adverse Events and SAE will be assessed by CTCAE5.0.
severity of TEAE and SAE | through study completion, an average of 6 months
  The Treatment-Related Adverse Events and SAE will be assessed by CTCAE5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gen Lin, Ph.D, Principal Investigator — Fujian Cancer Hospital

IPD SHARING:
Plan to Share IPD: No
Will decided after the study initiated.